CLINICAL TRIAL: NCT07245901
Title: An Investigator-initiated, Open-Label Clinical Study of a mRNA Vaccine Encoding Tumor-Specific Circular RNA Antigens in Combination With Anti-PD-1 Monoclonal Antibody in Patients With Advanced Solid Tumors
Brief Title: Safety and Tolerability of a mRNA Vaccine Encoding Tumor-Specific Circular RNA Antigens in Combination With Anti-PD-1 Monoclonal Antibody in Patients With Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Zenith Institute of Medical Sciences, Guangzhou (Unknown)
Responsible Party: Principal Investigator, Erwei Song, M.D., Ph.D., Ph.D, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2025-591-02
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-10

CONDITIONS: Solid Tumor
Keywords: Tumor vaccine; mRNA vaccine; solid tumor; immunotherapy
MeSH Terms: interventions — toripalimab; spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose Escalation phase (Experimental): A single dose of the PD-1 monoclonal antibody will be administered first, followed by combination treatment with the mRNA vaccine and the PD-1 antibody 21 days later. Participants will receive circFAM53B mRNA injection via an intramuscular (IM) injection on Day 1 of each 21-day cycle for up to 9 cycles, combined with PD-1 monoclonal antibody therapy for up to 35 cycles.
  Interventions: Drug: circFAM53B mRNA vaccine; Drug: toripalimab
- Dose Expansion phase (Experimental): A single dose of the PD-1 monoclonal antibody will be administered first, followed by combination treatment with the mRNA vaccine and the PD-1 antibody 21 days later. Participants will receive circFAM53B mRNA injection via an intramuscular (IM) injection on Day 1 of each 21-day cycle for up to 9 cycles, combined with PD-1 monoclonal antibody therapy for up to 35 cycles.
  Interventions: Drug: circFAM53B mRNA vaccine; Drug: toripalimab

INTERVENTIONS:
Drug: circFAM53B mRNA vaccine — IM injection on Day 1 of each 21-day cycle for up to 9 cycles
  Other Names: circFAM53B mRNA injection
Drug: toripalimab — Intravenous infusion once every 21 days
  Other Names: anti-PD-1 monoclonal antibody

SUMMARY:
This is an Investigator-initiated, Open-Label Clinical Study of a mRNA Vaccine Encoding Tumor-Specific Circular RNA Antigens in Combination with anti-PD-1 monoclonal antibody in Patients with Advanced Solid Tumors. Preclinical studies of this project have identified that circFAM53B, which is specifically overexpressed in tumor cells, possesses the ability to encode a cryptic peptide, FAM53B-219aa, representing a potential tumor vaccine target. In this study, the sequence encoding the cryptic antigen from circFAM53B will be linearized and formulated as an mRNA vaccine (circFAM53B mRNA injection). The vaccine will be administered via lipid nanoparticle (LNP) encapsulation, and its safety and efficacy will be evaluated in combination with anti-PD-1 monoclonal antibody therapy.

DETAILED DESCRIPTION:
This investigator-initiated clinical trial is designed to evaluate the safety and preliminary efficacy of the circFAM53B mRNA vaccine in combination with anti-PD-1 monoclonal antibody therapy using a "3+3" dose-escalation design. The trial consists of two phases: a dose-escalation phase and a dose-expansion phase.

In the dose-escalation phase, patients with advanced solid tumors exhibiting high circFAM53B-219aa expression who have failed prior standard therapies will be enrolled. Approximately 10-20 participants will receive the circFAM53B mRNA vaccine to determine the safety profile (DLT) and identify the maximum tolerated dose (MTD).

Based on the results from the dose-escalation phase, the dose-expansion phase will be conducted at the identified MTD. This phase will enroll participants from two different tumor types, with approximately 10 patients per cohort, to receive the circFAM53B mRNA vaccine in combination with toripalimab.

ELIGIBILITY:
Inclusion Criteria:

Voluntary participation: The patient voluntarily agrees to participate in the study, signs a written informed consent form (ICF), and is willing and able to comply with the study protocol requirements.

Age and sex: Male or female patients aged ≥18 years.

Life expectancy: Expected survival of ≥3 months.

Diagnosis: Histologically or cytologically confirmed unresectable or metastatic advanced solid malignancies, including but not limited to pancreatic cancer, breast cancer, non-small cell lung cancer, melanoma, and colorectal cancer.

Tumor tissue availability: Patients must have adequate fresh tumor tissue obtained via biopsy or surgery prior to treatment, or available formalin-fixed paraffin-embedded (FFPE) samples. The expression of circFAM53B-219aa in the specimen must be confirmed by RT-qPCR analysis and/or immunohistochemistry.

HLA genotyping will be performed using peripheral blood samples, employing polymerase chain reaction-sequence-based typing (PCR-SBT) combined with Sanger sequencing, with allele assignment referenced to the IMGT/HLA database, or alternatively, using PCR with sequence-specific oligonucleotide (SSO) probes, sequence-specific primers (SSP), or next-generation sequencing (NGS) technologies. Subsequently, NetMHCpan and MHCflurry predictive models will be applied to identify tumor-specific circFAM53B-39aa-derived peptides that bind to HLA class I molecules (HLA-A, -B, and -C) and to evaluate their binding affinity. Patients with HLA genotypes showing a predicted binding rank value <2 will be eligible for enrollment.

Measurable disease: At least one measurable lesion or bone-only lesion as defined by RECIST v1.1 (see Appendix 4: Response Evaluation Criteria in Solid Tumors).

Prior therapy: Patients who have failed standard therapy, have no available standard treatment, or cannot tolerate standard treatment-related toxicities.

Performance status: ECOG performance status 0-2.

Adequate organ function as defined below:

1. Hematology:

   * Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L;
   * Platelet count (PLT) ≥ 75 × 10⁹/L;
   * Hemoglobin (Hb) ≥ 90 g/L.
2. Hepatic function:

   • AST, ALT, and alkaline phosphatase ≤ 2.5 × ULN; total bilirubin (TBIL) ≤ 1.5 × ULN.

   Exceptions:
   * Patients with confirmed liver metastases: AST and/or ALT ≤ 5 × ULN;
   * Patients with confirmed liver or bone metastases: alkaline phosphatase ≤ 5 × ULN;
   * Patients with confirmed Gilbert's syndrome: total bilirubin ≤ 3.0 mg/dL.
3. Renal function: Serum creatinine ≤ 1.5 × ULN.
4. Coagulation: APTT ≤ 1.5 × ULN, and INR or PT ≤ 1.5 × ULN.
5. Cardiac function: Left ventricular ejection fraction (LVEF) ≥ 50% by echocardiography.
6. Pulmonary function: FEV₁ ≥ 60%.

Contraception: Fertile patients who are not surgically sterile must agree to use at least one medically approved contraceptive method (e.g., intrauterine device, oral contraceptives, or condoms) during the study treatment period and for 1 year after study completion. Female patients of childbearing potential must have a negative serum hCG test within 7 days prior to cell injection.

Recovery from prior therapy: Any toxicities from previous treatments must have resolved to CTCAE v5.0 Grade ≤1 or met protocol-specified laboratory criteria, except for:

Grade 2 peripheral neuropathy, alopecia, or vitiligo;

Hypothyroidism controlled with hormone replacement therapy;

Type I diabetes well controlled with insulin;

Other irreversible toxicities deemed by the investigator unlikely to worsen with vaccination.

Exclusion Criteria:

Participants meeting any of the following criteria will be excluded from the study:

Active infection requiring systemic therapy.

Uncontrolled tumor-associated pain, as determined by the investigator. Patients requiring analgesic therapy must be on a stable pain management regimen prior to enrollment. Symptomatic lesions amenable to palliative radiotherapy should be treated before study entry.

Severe cardiac disease or cardiac dysfunction expected to preclude tolerance to treatment, including but not limited to: life-threatening arrhythmias or high-grade atrioventricular block, unstable angina, clinically significant valvular heart disease, electrocardiographic evidence of transmural myocardial infarction, or uncontrolled hypertension.

Receipt of radiotherapy, chemotherapy, or endocrine therapy within 4 weeks prior to enrollment, or current participation in another interventional clinical trial.

Pregnant or breastfeeding women.

Active autoimmune disease, a history of autoimmune disease, or conditions requiring systemic corticosteroids or immunosuppressive therapy (>10 mg/day prednisone or equivalent).

Exceptions: hormone replacement therapy (e.g., thyroxine, insulin, or physiological corticosteroid replacement for adrenal or pituitary insufficiency) is permitted.

History of congenital or acquired immunodeficiency, including HIV seropositivity.

Active tuberculosis (TB) infection within 1 year prior to enrollment, or a history of active TB infection more than 1 year ago that was not adequately treated.

Active hepatitis B or C infection.

Patients who are HBsAg or HBcAb positive may be enrolled if HBV DNA is below the lower limit of normal (LLN) at the study site.

Patients who are HCV antibody positive may be enrolled if HCV RNA is below the LLN at the study site.

Carriers participating in the study should receive antiviral therapy as appropriate, with periodic quantitative nucleic acid testing during the study.

Active syphilis.

Receipt of any form of vaccination within 4 weeks prior to enrollment, or planned vaccination during the study period.

Previous allogeneic bone marrow transplantation or solid organ transplantation.

History of hypersensitivity or allergic reactions to any component of the investigational products, including but not limited to the mRNA vaccine, toripalimab, or their formulation excipients.

Concurrent use of prohibited concomitant medications, such as systemic corticosteroids or live vaccines, unless discontinued at least 7 days prior to enrollment.

Any other condition that, in the investigator's judgment, may compromise patient safety, treatment compliance, or study integrity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-05 (Estimated); Primary Completion 2028-12-05 (Estimated); Study Completion 2030-12-05 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | 12 months
  Safety and tolerability as determined by assessment of dose limiting toxicities and the maximum tolerated dose or maximal assessed dose per protocol of the vaccine with cancers.
Recommended Phase 2 Dose (RP2D) | 12 months
  To determine a recommended phase 2 dose of the vaccine for further development by evaluating number of patients with treatment-related adverse events as assessed by the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0)
Maximum Tolerated Dose (MTD) | 12 months
  Determine the maximum tolerated dose by assessing the Incidence of Dose Limiting Toxicities (DLTs), treatment emergent and treatment related adverse events (assessed by CTCAE v5.0).

SECONDARY OUTCOMES:
Overall Response Rate (ORR): Number of Participants with Tumor Response (Partial or Complete) | Baseline through disease progression by Response Evaluation Criteria of Solid Tumors Version 1.1 (RECIST 1.1), start of new anti-cancer therapy, withdrawal of consent, death and last safety follow-up visit (up to approximately 3 years)
  ORR is defined as the proportion of participants whose best overall response is complete response (CR) or partial response (PR).
Duration of Response (DoR) | Baseline through disease progression by RECIST 1.1, start of new anti-cancer therapy, withdrawal of consent, death and last safety follow-up visit (up to approximately 3 years)
  DoR is defined as time from first tumor response (partial or complete) until either radiological disease progression, clinical/symptomatic disease progression or death (whichever is sooner).
Progression Free Survival (PFS) | Baseline through disease progression by RECIST 1.1, start of new anti-cancer therapy, withdrawal of consent, death and last safety follow-up visit (up to approximately 3 years)
  PFS is defined as time between the date of first dose of Toripalimab and the date of either radiological disease progression, clinical/symptomatic disease progression or death (whichever is sooner).
Overall Survival (OS) | Baseline to death of any cause (up to approximately 3 years)
  OS is defined as time between the date of the first dose of study drug and the date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Erwei Song, Study Chair — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University

IPD SHARING:
Plan to Share IPD: No